CLINICAL TRIAL: NCT01596907
Title: Treatment of Low Metabolic Rate and Low Weight Loss Rate Following Bariatric Surgery
Brief Title: Treatment of Low Metabolic Rate Following Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Weight Loss Surgery, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 115183
Record Dates: First submitted 2012-05-08; First posted 2012-05-11 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Morbid Obesity
Keywords: resting energy expenditure; fat free mass; lean body mass; bariatric surgery; morbid obesity; ephedrine; caffeine; Low metabolic rate; Low lean body mass; Weight loss rate
MeSH Terms: conditions — Obesity, Morbid | interventions — Ephedrine; Caffeine; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ephedrine and caffiene (Active Comparator): Drug treatment:
  ephedrine sulfate 25-mg with caffeine 200-mg per capsule to be given three times per day 4 hours apart for 6 months after gastric bypass surgery. Weight loss rate, resting energy expenditure, fat free mass will be measured during the treatment.
  Interventions: Drug: Ephedrine sulfate with caffeine
- placebo (Placebo Comparator): one placebo capsule will be taken three times per day 4 hours apart, identical to the instructions for the active drug for approximately 6 months following gastric bypass surgery. Weight loss rate, resting energy expenditure and fat free mass will be measured during the treatment.
  Interventions: Drug: cellulose

INTERVENTIONS:
Drug: Ephedrine sulfate with caffeine — Ephedrine sulfate 25-mg with caffeine 200-mg combination capsule to start 5 weeks after gastric bypass surgery at 3 times per day 4 hours apart.
  Arms: Ephedrine and caffiene
Drug: cellulose — sufficient cellulose to fill a placebo capsule identical to the active drug to be taken 3 times per day 4 hours apart for 6 months after gastric bypass surgery
  Arms: placebo

SUMMARY:
Purpose is to determine the effect of ephedrine and caffeine, on metabolic rate and weight loss after bariatric surgery. Approximately 40% of patients struggle with their weight loss rate, or metabolic rate, after bariatric surgery, and at least 30% previously had or develop a low metabolic rate after surgery. Metabolic rate is the speed at which calories are burned. The fewer the calories eaten and the more calories burned, the more rapidly weight is lost. It is possible that despite a very low calorie intake following bariatric surgery metabolic rate will decrease so much so that weight does not decrease even if intake is reduced to 1000 calories per day. Ephedrine is a medicine used commonly to treat asthma, difficulty breathing, and wheezing. However, 40 years ago it was reported in scientific studies that ephedrine increases weight loss in patients on low calorie diets by increase the amount of calories that are burned. Combining caffeine with ephedrine makes ephedrine work more efficiently (more weight loss over time). Many studies show the effect of ephedrine on weight loss that began in 1974 with patients on food diets. Ephedrine used in various strengths and with a number of different combinations has shown to be effective and safe, especially when directed by a physician. There is only one study where ephedrine has been used in patients after bariatric surgery. In that study, both the patient and medical staff knew they were taking ephedrine (i.e., they were not "blinded"). The patients who were not losing weight or had measured low metabolic rates were treated with ephedrine. The patients taking ephedrine lost more weight after surgery than those not taking ephedrine. While this is a significant finding, the study was not designed to be the best test of the effects of ephedrine. The best test is where neither the patients nor the medical staff know if the patient is taking the active drug (double blind). All patients enrolled into the Research Study will receive capsules that contain either ephedrine and caffeine (the active drug) or identical capsules with no active ingredient (called a "placebo"). Neither group of patients will know which set of capsules they receive. The expected duration of treatment in the Study is 7 months from the day of surgery. This is a single site study. All patients will have their gastric bypass performed through Oregon Weight Loss Surgery at Legacy Good Samaritan Hospital. The investigators expect to study 200 patients with 100 receiving the study drugs (ephedrine and caffeine in a capsule) and 100 receiving placebo (inactive ingredients in an identical capsule) over approximately 6 months.

DETAILED DESCRIPTION:
Research Objectives:

The primary objective is to apply an effective medical weight loss treatment to post bariatric surgery patients to enhance their weight loss through stimulation of thermogenesis and lipolysis and retention of lean body mass. This treatment using ephedrine with phosphodiesterase inhibitor (caffeine or theophylline) has been extensively documented as safe and effective in the medical weight loss setting but has not been applied to post-bariatric surgery patients in a placebo controlled, double blind, randomized study. From preliminary studies this treatment should be effective, especially in the treatment of post-surgical patients who continue to have difficulty losing weight despite good activity levels and significant calorie restriction.

Clinical Relevance:

Raum and others have been treating patients presenting with low metabolic rates during medical and bariatric surgery induced weight loss for many years with ephedrine in combination with caffeine and/or theophylline. All the literature outlined below for the last 40 years have been conducted only during medical weight loss. There are no randomized trials in surgical patients. Abstracts and expert opinion papers have been published but without randomization or blinding.

Ephedrine has become controversial despite considerable evidence of its safe and effective treatment of airway resistance (asthma) for 50 years, and its use for medical weight loss (to stimulate REE and prevent loss of lean body mass) since 1974. An association with a non-regulated food additive, ephedra sparked the initial problems with inappropriate dosing, lack of physician supervision for patient selection and sensationalism in the lay press unsupported by peer-reviewed studies to contradict previous favorable studies. Secondly, using ephedrine and pseudoephedrine as substrate for the illegal manufacture of methamphetamine, caused an aura of further unreasoned apprehension. Because ephedrine with caffeine or theophylline is one of the few drug combinations that can potentially reverse a low REE and allow a successful weight loss following bariatric surgery, a randomized, controlled study is needed to determine if this effect is statistically and clinically significant in patients having bariatric surgery.

SPECIFIC AIMS Background and Current Research Following bariatric surgery, metabolic rate decreases secondary to a decrease in sympathetic activity and lean body mass preventing optimal weight loss (1-3). Patients reaching this "plateau" during weight loss be it medical or surgical is well recognized. The plateau is reached when there is no longer a significant difference between calories burned and calories consumed. The equation can be modified at either end. High calorie intake is, by far, the most common reason given for lack of weight loss. The advice provided is to decrease calorie intake. However, there is a large subgroup of individuals whose metabolic rate (measured as Resting Energy Expenditure - REE or Resting Metabolic Rate - RMR) decreases while caloric intake has remained low. Raum (3) has routinely measured REE in bariatric surgery patients for 10 years. A low REE is commonly associated with a reduced weight loss rate. Hundreds of patients have been found to have REEs significantly depressed from normal (90-s100%) to a range of 45% to 80% and a mean of 65%. These patients have a deficit of 500 to more than 1000 kcal per day that they would be burning with a normal REE. Some patients must consume less than 700 to 1000 kcal/day just to maintain their weight.

The methods to increase REE, sympathetic activity, brown adipose tissue activity include exercise, and several drugs including catechins (green tea), caffeine or theophylline with ephedrine, and capsaicin (1). Many clinical trials have demonstrated the effect of ephedrine on weight loss (4-7). A significant effect of ephedrine on increasing metabolism is thought to be one of the mechanisms for weight loss. Stimulation of brown adipose tissue was thought to contribute to 15% of the increase in thermogenesis and the remainder due to thermogenesis in muscle (8). Combinations of ephedrine with methylxanthines (caffeine and/or theophylline) are noted to be even more effective in raising metabolic rates. These effects were most notable in post-obese patients who had some lost some weight, and had depressed metabolic rates. REE increased 8% in the post-obese but had no effect in lean subjects. In the previously obese subjects, the ephedrine-methylxanthine combination normalized the defective thermogenic response to a meal (9). In a 24-week trial with 20 mg of ephedrine and 200 mg of caffeine tid were randomized with placebo. The ephedrine/caffeine group lost 17.5% of body weight with 25% of the weight loss attributed to thermogenesis (10). The thermogenic effect of ephedrine may be lost early in treatment but is restored with the addition of aminophylline (11).

The effect of ephedrine on body composition has been studied. Two groups were given a very low calorie diet. Placebo or Ephedrine in combinations with or without methylxanthines and/or aspirin (110 mg tid) in an 8 week trial demonstrated no side effects. The ephedrine groups lost 4.5 kg more fat and 2.5 kg less lean than the placebo, significant differences. REE fell 13% in the placebo group, but only 8% in the ephedrine groups (18).

A few examples of the literature were highlighted above that reflect similar studies that can be found in extensive reviews of ephedrine on weight loss (19-26), energy balance and thermogenesis (27,28).

Considerable recent controversy about the safety of ephedrine has come to pass due to the widespread use of an herbal food additive, ephedra, being marketed widely beginning in the late 1990s. Ephedrine had been used without controversy from the 1960s until this time. Many anecdotal reports were circulated, including over 18,000 case reports. These and 550 trials were reviewed in a meta-analysis (30). Of these reports less than 10% of the trials could be scientifically assessed and of these only 22 consisted of a placebo with some combination of ephedrine, ephedra, caffeine or other herbs. These remaining studies demonstrated a 2.2 to 3.6 fold increase in one or more of the following grouped subjective complaints, psychological, gastrointestinal, autonomic symptoms, and/or palpitations. Presumably the other 90% of actual trials did not test or did not highlight these symptoms. Other papers (31-33) which were reviews of various types of reports (not designed studies) described instances of acute intoxication resulting in strokes, heart attacks, seizure and even death. Because of the uncontrolled nature of the data in the reports, doses, combinations with other drugs, and frequency or duration of exposure were unknown, they could only state whether the associations with ephedra were possible or probable.

Other research observed no significant adverse effects or only temporary minor effects with ephedra, ephedrine and caffeine (13, 14, 34-37). These studies were double-blind placebo controlled in selected populations. Multiple clinical weight loss trials have measured the chronic and acute effects of combinations of ephedrine (30, 60 and 150 mg per day) with caffeine (300 to 600 mg per day) up to 180 subjects over 24 weeks (10, 12-15). Acutely, mean arterial pressure is increased by 9 mm/Hg and pulse by 7 beats per minute. By 8 weeks the side effects of tremor, insomnia, dizziness and blood pressure initially noted with ephedrine were equal to placebo. In some studies side effects were only seen at the highest dose of 50 mg tid (16). No adverse effects were noted with a dose of ephedrine 25 mg and caffeine 200 mg tid for 10 days on cardiovascular function as measured by thoracic bio-impedance, automatic sphygmomanometry, continuous electrocardiographic recording or ergometric exercise (17).

The difference between these two contrasting sets of data demonstrates that the unregulated use of ephedrine-containing compounds in unknown and potentially lethal doses in susceptible populations is not to be encouraged. But in preparations where dosage is known and controlled, given in appropriately selected populations, ephedrine with caffeine is safe and effective.

References available on request.

EXPERIMENTAL STUDY DESIGN Patients who have been medically cleared for gastric bypass surgery and meet the inclusion criteria or are not eliminated by the exclusion criteria will be offered the opportunity to enroll in the study.

Patients will be enrolled in the study, IRB consents obtained, and randomized to treatment or control groups prior to surgery. Patients will follow all usual preoperative and postoperative surgical and medical investigations and care. This includes a baseline resting energy expenditure (REE) and body composition measurement (BC) before surgery. Study visits will usually occur at the same times as normal follow up visits and vital signs and weights obtained.

Patients will begin taking ephedrine/caffeine or placebo capsules at 5 weeks after surgery in a gradual tapering dose upward beginning with one capsule daily and increasing each week by one capsule until taking three capsules per day. For the treatment group this would be 75 mg of ephedrine and 600 mg of caffeine per day. At 8 weeks after surgery they will return for an office visit, vital signs taken, BC done, symptom checklist completed and reviewed, and if not experiencing any significant side effects they will be given a 6 weeks supply of capsules. At 14 weeks after surgery they have and office visit with vital signs taken, symptom checklist completed and reviewed and be given another 6 week supply of capsules. At 20 weeks after surgery they have and office visit with vital signs taken, symptom checklist completed and reviewed, and an REE study will be obtained at Good Samaritan hospital and body composition by bioimpedance in the clinic and be given another 6 week supply of capsules. At 26 weeks after surgery they have and office visit with vital signs taken, symptom checklist completed and reviewed and be given another 6 week supply of capsules. At 32 weeks after surgery they will return for an office visit for vital signs, a symptom checklist and an REE study will be obtained at Good Samaritan hospital and body composition by bioimpedance in the clinic. They will be given a taper pack of capsules that will be accomplished over 3 weeks.

At the clinic visits noted above vital signs, and body weight will be obtained. Patients will be questioned about any side effects. They will also be encouraged to call between visits if they have persistent side effects, and will be given a symptom checklist to compare over the phone. As usual routine medical and surgical care will be provided at these visits. Adjustments in medications for blood pressure, diabetes, hyperlipidemia, nutritional deficiencies and so forth will be addressed and treated as usual. Any surgical interventions for wound problems, hernias, or other complications will be attended to and routine blood tests or any other diagnostic tests needed, will be done. If blood pressure cannot be controlled to < 140/80, or pulse < 100, or patient experiences excessive adrenergic side effects, the treatment will be stopped, but the patient will continue with usual follow up medical and surgical care. The investigators will continue to collect measurements on patients who are unable to tolerate the treatment until the end of the study. Patients may withdraw, however, at anytime without any repercussions and will continue to receive regular care.

Body composition will be measured by body impedance analysis with a Quantum III BIA from RJL Systems (Michigan). This is a high quality, reproducible system using electrode placement on hands and feet. While DEXA body scans may provide more detailed information the research cost for these measurements in this study would exceed the cost of the medications alone. The investigators have three RJL systems in the clinic and the total body lean mass compares well the comparable measurements obtained with the DEXA.

REE is measured using a Sensor Medics indirect calorimeter with O2 and CO2 measurements to calculate REE. This equipment is located and managed by the Respiratory Therapy Department at Good Samaritan Hospital and has been calibrated, tested and used in other funded research studies. The test is done fasting, without morning medications with minimal pretest activity (15 minutes at rest prior to starting the test), and normal fluid balance. The equipment is calibrated before each test.

Body weights are obtained on an electronic scale, capacity 800 pounds, with shoes off and patients are advised to wear the same light weight clothes at each visit. The scale's calibration is checked quarterly (a requirement of current and prior research studies).

The investigators use a Welch-Allyn automatic cuff for blood pressure and pulse. Two measurements are obtained in each arm at each visit. The investigators have multiple size cuffs to match upper arm diameter. Calibration checked quarterly as research protocols have required.

Power analysis was performed with results from our previous studies in non-randomized subjects treated for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Qualify for gastric bypass or sleeve gastrectomy (fertile females with negative pregnancy test)
* Willing to comply with scheduled follow up appointments
* Blood pressure < 140/80 and heart rate < 100 measured three times

Exclusion Criteria:

* Treated hypertension with blood pressure still > 140/80
* Stroke or myocardial infarction within the last 12 months
* Angina currently requiring medical treatment
* On medication or a device to control arrhythmias
* On a beta blocker to treat hypertension
* On medications known to interact with ephedrine or caffeine
* Unable to tolerate side effects
* Pregnancy
* Fertile females unwilling to practice effective birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Resting Energy Expenditure from baseline | 3 and 6 months after treatment begins
  By indirect calorimetry resting energy expenditure will be calculated from vO2 and vCO2 ratios using the Harris-Benedict Equations
Change in Body Composition from baseline | 3 months and 6 months after beginning treatment
  Body Impedance Analysis will be measured at each office visit before and after beginning treatment using a Quantum III BIA from RJL Systems (Michigan)

SECONDARY OUTCOMES:
Change in Body Mass Index from baseline | 8, 14, 20, 26, 32 weeks after treatment
  Body Mass Index will be calculated from weight and height obtained at each office visit.
Arterial Blood Pressure | 8, 14, 20, 26, 32 weeks after treatment
  Arterial blood pressure will be obtain in both arms times two at each office visit.
Heart Rate | 8, 14, 20, 26, 32 weeks after treatment
  Heart rate will be determined at two time points in each arm at each office visit.

CONTACTS AND LOCATIONS:
Overall Officials: William J Raum, MD PhD, Principal Investigator — Oregon Weight Loss Surgery
Locations (2):
- United States (2):
  - Oregon Weight Loss Surgery, LLC, Beaverton, Oregon
  - Oregon Weight Loss Surgery, Portland, Oregon